CLINICAL TRIAL: NCT04963192
Title: Integrated Management of Chronic Respiratory Diseases - eMEUSE-SANTE
Brief Title: Integrated Management of Chronic Respiratory Diseases
Acronym: eMEUSE-SANTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: EFCR Department and Sleep Laboratory, Grenoble Alpes University Hospital (Unknown); Pneumology Department, Verdun Hospital (Unknown); BIOSENCY compagny (Unknown); SEFAM compagnie (Unknown); ADOR - Territorial Support Network, Device and Tools for Primary Care Teams (Unknown); PULSY - Regional Support Group for the Development of e-health (Unknown); eMeuse-Santé consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A01126-35; 38RC21.149 (Other: Grenoble Alpes University Hospital)
Record Dates: First submitted 2021-06-21; First posted 2021-07-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Sleep Apnea, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A prospective clinical study, conducted at the Verdun Hospital, in patients with a chronic respiratory pathology (OSA or COPD), including an integrated management at home using connected devices, during 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSA or COPD patients having an integrated management at home (Experimental): OSA or COPD patients having an integrated management at home using connected devices, during 6 months
  Interventions: Device: Connected actimeter to measure physical activity in OSA patients; Device: Connected BORA Band to measure physical activity in COPD patients only; Other: IPAQ to evaluated physical activity; Device: Connected scale to measure weight; Device: Connected tensiometer to measure arterial pressure; Device: Connected BORA Band to measure oxygen saturation in COPD patients only; Device: Connected BORA Band to measure heart rate in COPD patients only; Device: Connected BORA Band to measure respiratory rate in COPD patients only; Other: EXASCORE to evaluated COPD severity; Other: Epworth scale to evaluate sleepiness; Other: Pichot scale to evaluate fatigue; Other: Usability questionnaire; Other: SF36 questionnaire

INTERVENTIONS:
Device: Connected actimeter to measure physical activity in OSA patients — Connected actimeter worn for one week before initiation of treatment, at M3 and at M6, to measure average daily steps for OSA patients
Device: Connected BORA Band to measure physical activity in COPD patients only — Connected BORA Band worn for one week before initiation of treatment, at M3 and at M6, to measure average daily steps for COPD patients only
Other: IPAQ to evaluated physical activity — Physical activity evaluated by IPAQ (International Physical Activity Questionnaire) at the inclusion, M3 and M6
Device: Connected scale to measure weight — Weight measured by a connected scale, before CPAP or NIV treatment, at M3 and M6
Device: Connected tensiometer to measure arterial pressure — Arterial pressure measured by a connected tensiometer, before CPAP or NIV treatment, at M3 and M6
Device: Connected BORA Band to measure oxygen saturation in COPD patients only — Daily oxygen saturation measured by the connected BORA Band for COPD patients only during 6 months
Device: Connected BORA Band to measure heart rate in COPD patients only — Daily heart rate measured by the connected BORA Band for COPD patients only during 6 months
Device: Connected BORA Band to measure respiratory rate in COPD patients only — Daily respiratory rate measured by the connected BORA Band for COPD patients only during 6 months
Other: EXASCORE to evaluated COPD severity — COPD severity evaluated by the EXASCORE questionnaire at inclusion, M3 and M6 for COPD patients only
Other: Epworth scale to evaluate sleepiness — Sleepiness evaluated by the Epworth scale at baseline, M3 and M6
Other: Pichot scale to evaluate fatigue — Fatigue evaluated by the Pichot scale at inclusion, M3 and M6
Other: Usability questionnaire — Subjective assessment of each device by means of usability questionnaire at M6
Other: SF36 questionnaire — Quality of life evaluated by the SF36 questionnaire at inclusion and M6

SUMMARY:
Chronic respiratory diseases such as obstructive sleep apnea syndrome (OSA) and chronic obstructive pulmonary disease (COPD) constitute a major public health problem, due to their high prevalence, but especially because of their cardiovascular and metabolic morbidity and mortality and the associated costs for the health system. The organization of long-term management of these diseases is now part of the e-health process, digital health with the use of massive "big data" generated by care and follow-up. Therapeutic patient education and the integration of connected objects will allow personalized therapeutic education support with interventions by local medical staff adapted to the needs of the patients.

This will also allow to objectify the effect of treatments such as continuous positive airway pressure (CPAP) for OSA or non-invasive ventilation (NIV) and/or oxygen therapy for COPD, not only on the prevention of respiratory decompensation but also on cardiovascular and metabolic risk factors which are major elements of the prognosis. This project will therefore make it possible to demonstrate the feasibility and to deploy a multi-actor care pathway in the territory.

The investigators propose a prospective clinical study, conducted at the Verdun Hospital, with the main objective of studying the evolution of the quality of life of patients with a chronic respiratory pathology, during an integrated management at home for 6 months.

The secondary objectives:

* To study the evolution of the following parameters, before treatment (at inclusion) and after 6 months of integrated management:

  1. Treatment compliance (CPAP or NIV/oxygen therapy)
  2. Physical activity
  3. Weight
  4. Mean arterial pressure
  5. Oxygen saturation, heart rate and respiratory rate for COPD patients
  6. Severity of COPD for the patients concerned
  7. Daytime sleepiness
  8. Fatigue
  9. Patient acceptability of the use of connected objects
* To analyze the trajectories of the measures collected throughout the integrated management to identify specific profiles.
* To analyze the daily data of the different connected objects and treatments with regard to the patients' profiles (according to age, gender, comorbidities, OSA or COPD group).

DETAILED DESCRIPTION:
Chronic respiratory diseases such as obstructive sleep apnea syndrome (OSA) and chronic obstructive pulmonary disease (COPD) constitute a major public health problem, due to their high prevalence, but especially because of their cardiovascular and metabolic morbidity and mortality and the associated costs for the health system. There is also an inequality of access to referral care linked to demographics and territorial organization. We are currently at a turning point in the understanding of these pathologies and their coordinated management by combining therapeutic modalities. The organization of long-term management of these diseases is now part of the e-health process, digital health with the use of massive "big data" generated by care and follow-up. Therapeutic patient education and the integration of connected objects measuring weight, oxygen saturation rate, heart rate, respiratory rate, skin temperature blood pressure or physical activity will allow personalized therapeutic education support with interventions by local medical staff adapted to the needs of the patients.

This will also allow to objectify the effect of treatments such as continuous positive airway pressure (CPAP) for OSA or non-invasive ventilation (NIV) and/or oxygen therapy for COPD, not only on the prevention of respiratory decompensation but also on cardiovascular and metabolic risk factors which are major elements of the prognosis. This project will therefore make it possible to demonstrate the feasibility and to deploy a multi-actor care pathway in the territory.

The investigators propose a prospective clinical study, conducted at the Verdun Hospital, with the main objective of studying the evolution of the quality of life of patients with a chronic respiratory pathology, during an integrated management at home for 6 months.

The secondary objectives:

* To study the evolution of the following parameters, before treatment (at inclusion) and after 6 months of integrated management:

  1. Treatment compliance (CPAP or NIV/oxygen therapy)
  2. Physical activity, measured by an actimeter for OSAS patients or by the BORA Band device for COPD patients, for one week and IPAQ
  3. Weight, measured by a connected scale
  4. Average blood pressure, measured by a connected blood pressure monitor
  5. Oxygen saturation, heart rate and respiratory rate measured by the BORA Band for COPD patients
  6. The severity of COPD by the EXASCORE questionnaire for the patients concerned
  7. Daytime sleepiness by the Epworth questionnaire
  8. Fatigue by the Pichot scale
  9. Patients' acceptability of the use of the connected objects by questionnaires of satisfaction of use at 6 months.
* To analyze the trajectories of the measures collected throughout the integrated management to identify specific profiles.
* To analyze the daily data of the different connected objects and treatments with regard to the patients' profiles (according to age, gender, comorbidities, OSA or COPD group).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a chronic respiratory pathology such as:
* Newly diagnosed OSA with indication for CPAP treatment
* And/or COPD with or without indication for NIV/oxygen therapy
* Have a smartphone (with Android or iOS) allowing the installation of applications for connected objects
* Be able to use a mobile application on a personal smartphone
* Person agreeing to the telemonitoring of CPAP or NIV/oxygen therapy compliance data by the healthcare provider
* Patient who has provided consent to participate in the study
* Person affiliated to the social security

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient unable to give consent to participate in the study
* Patient under guardianship or curatorship
* Patient not affiliated to the social security system
* Patient deprived of liberty or hospitalized
* Patient protected by law
* Patient under administrative or judicial control
* Patient currently participating in another clinical research study that may have an impact on the study, this impact is left to the discretion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of Quality of life assessed by the SF36 questionnaire | at inclusion and at 6 months
  Change of quality of life, assessed by the SF36 questionnaire, from Baseline (at inclusion) and after 6 months of an integrated management at home

SECONDARY OUTCOMES:
Change of Physical activity (average daily steps) for OSA patient only | One week before initiation of CPAP treatment and at Month 3 and Month 6
  Change of the physical activity using a connected actimeter for OSA patients only, from Baseline (one week before treatment) and after 3 and 6 months of an integrated management at home
Change of Physical activity (average daily steps) for COPD patient only | One week before initiation of NIV treatment and at Month 3 and Month 6
  Change of the physical activity using the connected BORA Band for COPD patients only, from Baseline (one week before treatment) and after 3 and 6 months of an integrated management at home
Change of Physical activity assessed by the IPAQ questionnaire | At the inclusion, Month 3 and Month 6
  Change of Physical activity assessed by the IPAQ (International Physical Activity Questionnaire), from Baseline (at inclusion) and after 3 and 6 months of an integrated management at home
Change of Weight measured by a connected scale | Before CPAP or NIV treatment, at Month 3 and Month 6
  Change of Weight measured by a connected scale, from Baseline (before CPAP or NIV treatment), and after 3 and 6 months of an integrated management at home.
Change of Arterial pressure measured by a connected tensiometer | Before CPAP or NIV treatment, at Month 3 and Month 6
  Change of Arterial pressure measured by a connected tensiometer, from Baseline (before CPAP or NIV treatment), and after 3 and 6 months of an integrated management at home.
Daily oxygen saturation measured by the connected BORA Band for COPD patients only | During 6 months
  Daily oxygen saturation measured by the connected BORA Band for COPD patients only
Daily heart rate measured by the connected BORA Band for COPD patients only | During 6 months
  Daily heart rate measured by the connected BORA Band for COPD patients only
Daily respiratory rate measured by the connected BORA Band for COPD patients only | During 6 months
  Daily respiratory rate measured by the connected BORA Band for COPD patients only
Change of COPD severity evaluated by the EXASCORE questionnaire for COPD patients only | At the inclusion, Month 3 and Month 6
  Change of COPD severity evaluated by the EXASCORE questionnaire for COPD patients only, from Baseline (at inclusion), and after 3 and 6 months of an integrated management at home.
Change of Sleepiness evaluated by the Epworth questionnaire | At baseline, Month 3 and Month 6
  Change of Sleepiness evaluated by the Epworth questionnaire, from Baseline (at inclusion), and after 3 and 6 months of an integrated management at home.
Change of Fatigue evaluated by the Pichot questionnaire | At inclusion, Month 3 and Month 6
  Change of Fatigue evaluated by the Pichot questionnaire, from Baseline (at inclusion), and after 3 and 6 months of an integrated management at home.
Satisfaction and usage of the connected scale assessed by a specific questionnaire | At Month 6
  Satisfaction and usage of the connected scale assessed by a specific questionnaire, after 6 months of an integrated management at home
Satisfaction and usage of the connected tensiometer assessed by a specific questionnaire | At Month 6
  Satisfaction and usage of the connected tensiometer assessed by a specific questionnaire, after 6 months of an integrated management at home
Satisfaction and usage of the connected actimeter assessed by a specific questionnaire, for OSA patients only | At Month 6
  Satisfaction and usage of the connected actimeter assessed by a specific questionnaire, for OSA patients only, after 6 months of an integrated management at home
Satisfaction and usage of the connected BORA Band assessed by a specific questionnaire, for COPD patients only | At Month 6
  Satisfaction and usage of the connected BORA Band assessed by a specific questionnaire, for COPD patients only, after 6 months of an integrated management at home

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (2):
- France (2):
  - Grenoble Alpes University Hospital, Grenoble
  - Verdun Hospital, Verdun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coiffier O, Bailly S, Joyeux-Faure M, Tamisier R, Amrani K, Cornu JC, Gentina T, Terrail R, Causse C, Lombardi C, Pengo MF, Parati G, Pepin JL. Home Blood Pressure Trajectories During 6 Months of Continuous Positive Airway Pressure Therapy: Results from the eMEUSE-SANTE and SLEEPCONNECT Clinic. Ann Am Thorac Soc. 2025 Sep 23. doi: 10.1513/AnnalsATS.202505-504OC. Online ahead of print. PMID 40986800